CLINICAL TRIAL: NCT01529619
Title: A 24-week, Open-label, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Rivastigmine Patch in Patients With Mild to Moderate Alzheimer's Disease (MMSE 10-23) Switched From Cholinesterase Inhibitors (Donepezil, Galantamine)
Brief Title: Efficacy, Safety and Tolerability of Rivastigmine Patch in Patients With Mild to Moderate Alzheimer's Disease Switched From Cholinesterase Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713D1403
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
Keywords: Rivastigmine; Alzheimer's disease; Transdermal patch
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- Rivastigmine 18 mg (Experimental): During the 16-week titration period patients received daily rivastigmine 4.5mg patch for the first 4 weeks, rivastigmine 9mg patch for the next 4 weeks, rivastigmine 13.5mg patch for the next 4 weeks and then rivastigmine 18mg patch for the final 4 weeks. For patients who experienced intolerability, the dose was adjusted downward. Patients then entered the 8-week maintenance period during which time they continued to receive the dose of rivastigmine they were taking at the end of the titration period.
  Interventions: Drug: Rivastigmine transdermal patch

INTERVENTIONS:
Drug: Rivastigmine transdermal patch

SUMMARY:
This is a multicenter study to evaluate the efficacy, safety and tolerability of Rivastigmine patch in patients with mild to moderate Alzheimer's disease switched from Cholinesterase Inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria
* A clinical diagnosis of probable AD according to NINCDS/ADRDA criteria
* An MMSE score of > or = 10 and < or = 23
* Continuous treatment with donepezil ≤ 5 mg/day or galantamine ≤ 24 mg/day for 4 weeks prior to baseline visit
* Patients having difficulties being treated orally with ChE inhibitors (donepezil or galantamine) as judged by the investigator. Difficulties are defined as:
* Inadequate compliance with the ChE inhibitors at screening and baseline
* Presence of caregiver's burden for administering drugs orally at screening and baseline
* Inadequate treatment (efficacious dose cannot be reached or inadequate compliance) with the ChE inhibitors because of adverse events at screening and baseline
* Patients with swallowing difficulties at screening and baseline

Exclusion Criteria:

* A current DSM-IV diagnosis of major depression
* Taken rivastigmine in the past
* A score of > 5 on the Modified Hachinski Ischemic Scale (MHIS)

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Alzheimer's Disease Assessment Scale - Japan Cognitive Subscale (ADAS-J cog) | Baseline and Week 24
  The Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) was used to measure change in cognitive function. The ADAS-J cog score ranges from 0-70, with higher total scores indicating more impairment. A negative change score indicates improvement from baseline.

SECONDARY OUTCOMES:
Adverse Events, Serious Adverse Events, Adverse event leading to discontinuation of study drug | Week 24
  Adverse Events: An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug.
Change From Baseline in Disability Assessment for Dementia (DAD) | Baseline and Week 24
  The Disability Assessment for Dementia (DAD) was used to assess levels of difficulty in activities of daily living (ADL). The DAD is administered through an interview with the caregiver. A total score is obtained by adding the rating for each question and converting this to a total score out of 100 (%). Higher scores represent less disability in ADL while lower scores indicate more dysfunction. A positive change score indicates an improvement from baseline.
Change From Baseline in Mini-Mental State Examination (MMSE) | Baseline and Week 24
  The MMSE is a screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement from baseline.
Change From Baseline in Japanese version of the Clinical global impression of change (J-CGIC) | Week 4, 8, 12, 16, 20, 24
  The J-CGIC is simple 7 grade investigator's impression scale (1. Markedly improved, 2. Improved, 3. Slightly improved, 4. No change, 5. Slightly aggravated, 6. Aggravated, 7. Markedly aggravated).
Change From Baseline in Modified Crichton Scale | Baseline and Week 4, 8, 12, 16, 20, 24
  Modified Crichton Scale that assess basic activation of daily living, communication functions, and quality of life The following 7 items will be evaluated by caregiver. Total score is in the 0 to 56 range. Higher score means more severe impairment.
  Orientation, Conversation, Cooperation with family and caregiver, Restlessness, Dressing and clothes, Job and social activities/roles, Leisure activities
Formulation usability questionnaire | Week 24
  The Formulation usability preference questionnaire had been used to compare the previous oral AD drugs versus the patch The caregiver selects one of the following answers (1. Very easy to use, 2. Easy to use, 3. No change, 4. Not easy to use, 5. Not easy to use at all, 6. Unknown). The reason for the answer should be recorded as possible.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Japan (10):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Miyoshi, Hiroshima
  - Novartis Investigative Site, Ohtake, Hiroshima
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto